CLINICAL TRIAL: NCT01916824
Title: Effects of Treatment on Decision-making in Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Boadie W. Dunlop, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00066705
Record Dates: First submitted 2013-08-03; First posted 2013-08-06 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Major Depressive Disorder; Healthy Controls
Keywords: depression; melancholia; treatment
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — Sertraline; Citalopram; Escitalopram; Paroxetine; Fluoxetine; Vilazodone Hydrochloride; Venlafaxine Hydrochloride; Desvenlafaxine Succinate; Duloxetine Hydrochloride; Bupropion; Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Participants with Major Depressive Disorder (Experimental): Persons with a primary diagnosis of Major Depressive Disorder who start taking any FDA-approved antidepressant prescribed within standard dose range for 6 weeks
  Interventions: Drug: Any FDA Approved Antidepressant
- Healthy Controls (No Intervention): Persons without a history of Major Depressive Disorder and without a current diagnosis of any mental illness

INTERVENTIONS:
Drug: Any FDA Approved Antidepressant — Any FDA-approved antidepressant prescribed within standard dose range to treat Major Depressive Disorder will be taken for 6 weeks. Psychiatric follow-up will be performed during the study participation. At the end of the study, these participants will receive assistance in transitioning their care to another provider, depending on their individual circumstances.
  Other Names: Sertraline, Zoloft; Citalopram, Celexa; Escitalopram, Lexapro; Paroxetine, Paxil; Fluoxetine, Prozac; Vilazodone, Viibryd; Venlafaxine XR, Effexor XR; Desvenlafaxine, Pristiq; Duloxetine, Cymbalta; Bupropion, Wellbutrin; Mirtazapine, Remeron
  Arms: Participants with Major Depressive Disorder

SUMMARY:
In this trial, fifty participants with current major depressive disorder who are not receiving an antidepressant medication and fifty healthy controls will complete questionnaires and computerized tasks to assess their decision-making styles. There will be three visits for depressed patients and two for healthy controls (the first and third visits). The first visit will involve interviews and questionnaires to assess the participant's level of depression, medical history and quality of life. Participants will then complete the decision-making tasks, and will earn between $5-40 based on their choices, in order to make the decisions on the computer tasks financially meaningful. At the completion of this visit, depressed patients will be prescribed an FDA-approved antidepressant, chosen in consultation with the treating psychiatrist. Patients will be responsible for paying for the prescription themselves. After two weeks on the medication, the patient will be seen for a follow-up visit to ensure tolerability of the medicine. After six weeks on the medicine, patients and healthy controls will return to repeat the questionnaires and the computer based decision-making tasks, and will again earn between $5-40 based on their performance.

DETAILED DESCRIPTION:
During episodes of depression patients with major depressive disorder (MDD) may make sub-optimal decisions based on exaggerated negative beliefs about themselves, the future, or the world around them. These disruptions in decision-making contribute adversely to quality of life, in both work and personal realms. Although effective treatments for depression are available, very little work has explored the effects of treatment on how people make decisions. The specific aspects of decision-making that differ between depressed and health control individuals are unknown, and whether any changes in these decision-making features occur as a result of improvement from depression, or whether medication treatment itself can lead to changes in decision-making, even in the absence of clinical improvement.

In this trial, fifty participants with current major depressive disorder who are not receiving an antidepressant medication and fifty healthy controls will complete questionnaires and computerized tasks to assess their decision-making styles. There will be three visits for depressed patients and two for healthy controls (the first and third visits). The first visit will involve interviews and questionnaires to assess the participant's level of depression, medical history and quality of life. Participants will then complete the decision-making tasks, and will earn between $5-40 based on their choices, in order to make the decisions on the computer tasks financially meaningful. At the completion of this visit, depressed patients will be prescribed an FDA-approved antidepressant, chosen in consultation with the treating psychiatrist. Patients will be responsible for paying for the prescription themselves. After two weeks on the medication, the patient will be seen for a follow-up visit to ensure tolerability of the medicine. After six weeks on the medicine, patients and healthy controls will return to repeat the questionnaires and the computer based decision-making tasks, and will again earn between $5-40 based on their performance.

The overall goal of this study will be to identify whether decision-making characteristics in people with major depression is affected by treatment, and whether depressed patients make decisions differently from healthy controls. A total of 4 decision-making tasks and one control task will be administered via computer to eligible subjects. The specific tasks are:

1. Risk Task - This task assesses tolerance of risk by having participants decide whether they wish to accept a specific dollar payout, or to play a lottery with an uncertain payout.
2. Balloon Analogue Risk Task - The participant is presented with a balloon and offered the chance to earn money by pumping the balloon up by clicking a button. Each click causes the balloon to incrementally inflate and money to be added to a counter up until some threshold, at which point the balloon is over inflated and explodes. Thus, each pump confers greater risk but also greater potential reward. If the participant chooses to cash-out prior to the balloon exploding then they collect the money earned for that trial, but if balloon explodes earnings for that trial are lost. Participants are not informed about the balloons breakpoints; the absence of this information allows for testing both participants' initial responses to the task and changes in responding as they gain experience with the task contingencies.
3. Temporal Discounting Task - Participants are initially asked to choose between taking an immediate reward now or a larger reward at some time in the future. Decisions for seven time points over a 10-year time frame are proposed. The task is then repeated using choices between immediate and delayed losses, based on the same seven time points. This task assesses the manner in which subjects value immediate outcomes compared to long-term consequences.
4. Ultimatum Game - The ultimatum game (UG) is a well-established game-theoretical paradigm commonly employed in behavioral economics to measure emotional reactions to unfair offers. In the UG, two subjects sequentially exchange real monetary amounts. Specifically, a proposer is provided with a sum of money by the experimenter ($10), and asked to share this amount of money with another player, the responder. The responder then decides whether to accept or reject the offer made by the proposer. If the responder accepts the offer, both players receive the respective amounts from the proposer's offer. If she rejects the offer made by the proposer, both players receive nothing ($0). This is best illustrated via the following two potential scenarios: 1. the proposer offers a fair split of $5 for himself and $5 for the responder. This is an offer that is typically accepted by a great majority of responders. 2. The proposer offers a split of $9 for himself and $1 for the responder. Such offers are commonly rejected by the majority of responders, despite incurring a financial loss of $1.
5. Continuous Performance Task - This task involves identifying patterns of numbers briefly displayed on a computer screen. This task will serve as a control variable for attention in analyzing the results of the decision-making tasks.

ELIGIBILITY:
Inclusion Criteria for MDD Subjects:

1. Male or female, age 18-65
2. Primary Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV TR) Diagnosis of Major Depressive Disorder.
3. Has a 17-item Hamilton depression rating scale (HDRS-17) score >=16.
4. Ability to visually read and understand English language
5. Not currently taking an antidepressant.
6. Women of reproductive potential must be willing to take a medically approved form of birth control throughout the duration of the study.

Inclusion Criteria for Healthy Control Subjects:

1. Male or female, age 18-65
2. No current DSM-IV TR diagnosis of a mental illness.
3. No lifetime history of Major Depressive Disorder or Dysthymia.
4. Has a 17-item Hamilton depression rating scale (HDRS-17) score ≤7.
5. Ability to visually read and understand English language
6. Not currently taking any psychoactive medication

Exclusion Criteria for all subjects:

1. Has met criteria at any time during their life for bipolar disorder, a primary psychotic disorder (e.g. schizophrenia), or dementia.
2. Meet criteria for substance abuse or dependence within three months of the screening visit.
3. Presents with a clinically significant suicide risk, as assessed by a study physician.
4. Presence of any unstable or central nervous system-related medical illness that would interfere with cognition or participation.
5. Women who are currently pregnant or lactating, or plan to become pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boadie W Dunlop, MD, Principal Investigator — Emory University
Locations (1):
- Emory Mood and Anxiety Disorders Program, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from the Emory Mood and Anxiety Disorders Program between August 2013 and December 2015.
Pre-assignment Details: A total of 55 individuals gave informed consent to participate in the study. Of these, 2 were screen failures, resulting in 53 who began the trial.
Period: Overall Study
Arm/Group | Participants With Major Depressive Disorder | Healthy Controls
Started | 24 | 29
Completed | 17 | 20
Not Completed | 7 | 9
Not completed — Lost to Follow-up | 3 | 6
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: All participants who consented to take part in the study and fulfilled all eligibility criteria are included in the baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Major Depressive Disorder | Healthy Controls | Total
Number analyzed (Participants) | 24 | 29 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (11.3) | 31.4 (9.6) | 37.92 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 13 | 20
  White | 15 | 14 | 29
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 29 | 53

OUTCOME MEASURES:

1. Primary Outcome: Money Earned
Description: Change in amount of money earned between baseline and after 6 weeks of antidepressant treatment is determined through a summary score from a variety of decision-making tasks. Participants received between $5 and $40 per visit, depending on the outcomes of the decisions made on the computerized tasks. Variable payment ensured that the decision-making tasks were approached realistically, as opposed to using hypothetical "points" that do not have meaning in the real world. Greater earnings indicate better financial decision-making.
  The specific tasks were:
  1. risk task
  2. balloon analogue risk task
  3. temporal discounting task
  4. ultimatum game
  5. continuous performance task
Time Frame: Baseline, Week 6
Population: The population at each time point includes the number of participants completing the each visit.
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Participants With Major Depressive Disorder | Healthy Controls
Number analyzed (Participants) | 24 | 29
US Dollars
  Baseline Visit | 23.2 (5.6) | 25.0 (5.6)
  After 6 Weeks of Treatment: number analyzed (Participants) | 17 | 20
  After 6 Weeks of Treatment | 20.5 (6.6) | 21.9 (5.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time each participant provided informed consent throughout the entire 6 week duration of study participation.
Arm/Group | Participants With Major Depressive Disorder | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/29
Other Adverse Events (participants affected / at risk) | 12/24 | 2/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Major Depressive Disorder (N=24) | Healthy Controls (N=29)
Headache (General disorders) | 5 (5) | 2 (2)
Insomnia (General disorders) | 4 (4) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes